CLINICAL TRIAL: NCT05903079
Title: Impact of the Placebo Effect on the Effects of Trancranial Direct Current Stimulation in Fibromyalgia:A Randomized Clinical Trial
Brief Title: Impact of the Placebo Effect on the Effects of Trancranial Direct Current Stimulation in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Professor, surgery departament, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20220596
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, tDCS, Placebo effect
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Parallel Group, Sham-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The researcher will receive equipment already programmed by a research assistant, so the researcher who will deliver the tDCS to perform stimulation will not know the programed stimulation. Patients will be instructed to discuss aspects of treatment with the respective investigator. Two independent evaluators who will not participate in the consultations where guidance on the use of tDCS will be provided will be trained to make outcome assessments in follow-up. Patients will not be aware of the type of intervention received, since the sham condition produces a stimulus, but no expected effects. In order to study the level of the blinding, at each moment of evaluation, the patient will be asked about the type of intervention that he / she believes to have received (active or simulated), and about the degree of safety in the response, using a standardized questionnaire. The blinding will be evaluated at the end of each treatment week by means of a standardized instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respondres placebo effect (Placebo Comparator): Braço: Comparador de placebo: responde ao efeito placebo Intervenção: 'Estimulação Transcraniana por Corrente Contínua - tDCS
  Os pacientes receberão tratamento de estimulação tDCS córtex motor primário (M1).
  De acordo com o sistema 10-20 EEG, o ânodo será colocado no F3 esquerdo e o cátodo no FP2 direito.
  A estimulação placebo utiliza uma corrente de 2 miliamperes durante os primeiros minutos, nos 10 min e nos 19 minutos.
  Interventions: Device: s-Tdcs
- No Respondres placebo effect (Active Comparator): Braço: Comparador de placebo: responde ao efeito placebo Intervenção: 'Estimulação Transcraniana por Corrente Contínua - tDCS
  Os pacientes receberão tratamento de estimulação tDCS córtex motor primário (M1).De acordo com o sistema 10-20 EEG, o ânodo será colocado no F3 esquerdo e o cátodo no FP2 direitol.
  A estimulação placebo utiliza uma corrente de 2 miliamperes durante os primeiros minutos, nos 10 min e nos 19 minutos
  Interventions: Device: s-Tdcs

INTERVENTIONS:
Device: s-Tdcs — In the sham condition, a 2 mA current is applied only during brief ramp-up and ramp-down periods at the beginning of the session and at predefined time points (10 and 19 minutes), without sustained stimulation.
  In the active condition, a continuous 2 mA current is delivered for 20 minutes.

SUMMARY:
Fibromyalgia (FM) is a syndrome characterized by generalized musculoskeletal pain, fatigue, non-restorative sleep, cognitive alterations, depressive and neurovegetative symptoms. Conventional pharmacological therapies are known to produce responses with little clinical impact in more than 50% of patients. Functional alterations of the motor cortex and its connections with subcortical structures have also been demonstrated in FM. Based on the above, the objective of this research is to identify subgroups of patients with greater potential for response to treatment with a view to advancing diagnosis and treatment. In this study, the therapeutic target will be transcranial direct current stimulation (tDCS) according to the potential of responsiveness to the placebo effect, with the precise location of the stimulation area by a neuronavigation system, with the objective of counter-regulating the processes dysfunctional factors responsible for triggering and maintaining FM symptoms. Therefore, this clinical trial aims to compare the effectiveness of anodal tDCS applied to the primary motor cortex (M1) compared to sham tDCS in FM, according to susceptibility to the placebo effect and serum endorphin levels.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic disease that affects more than five million people annually in the US. The population prevalence ranges from 2% to 5.4% according to the 2010 American Society of Rheumatology diagnostic criteria. The female: male ratio has changed according to the diagnostic criteria. When applying the 1990 diagnostic criteria (ACR 1990) it is 7:1 and according to the 2010 criteria (ACR 2010) and revised in 2016, this ratio is 2.3:1. Regardless of the variation in prevalence between the sexes, it is a syndrome characterized by generalized musculoskeletal pain, fatigue, non-restorative sleep, cognitive changes, depressive symptoms and other correlates of autonomic dysfunction, such as colon syndrome. irritability and bladder tenesmus. In addition, FM has a level of psychological distress associated with catastrophism and depressive symptoms, which can worsen the prognosis and reinforce disability more markedly than is observed in other chronic pain conditions. FM is the prototype of dysfunction syndromes that course with pain by processes mediated by the central and peripheral nervous system. Patients with FM have been associated with an increased risk of stroke. In fact, it is a syndrome with great social impact, which demands advances in the understanding of diagnostic and therapeutic processes. In this direction, an attempt has been made to identify factors associated with the potential for response to treatment: potential for response to placebo, clinical, psychological, neurophysiological factors, levels of endorphins and neurotrophins associated with clinical response. The quest to understand the effects of these markers aims to personalize therapy and identify factors that can modify the clinical effect of treatments and the organization of neurobiological systems.

Although the results with the use of tDCS have been promising in the treatment of several chronic pain conditions, as demonstrated in a recent meta-analysis conducted by the Pain and Neuromodulation research group at Hospital de Clínicas de Porto Alegre (Zortea et al., 2019). ) it is necessary to consider that expectations about pain can directly affect nociceptive processing. Such expectations contribute to the placebo effect that has been shown to be mediated by opioids. The study by Eippert et al. (2009) showed that naloxone administration reduces the neural and behavioral effects of placebo, as well as placebo-induced responses in several cortical and subcortical areas that constitute the descending pain modulatory system (e.g., rACC, PAG, RVM, and hypothalamus). ). Furthermore, it abolished the rACC-PAG coupling induced by the placebo intervention. The expectation of placebo-induced analgesia is positively correlated with the availability of MOR. On the contrary, negative suggestion reduces the analgesic effects of synthetic opiates. All these findings support the close association between opioids and expectations that drive placebo-mediated analgesia.

Therefore, this clinical trial aims to compare the effectiveness of anodal tDCS applied to the primary motor cortex (M1) compared to sham tDCS in FM, according to susceptibility to the placebo effect and serum endorphin levels, in the following results ( 1) treatment efficacy, which includes daily measurements recorded in a Brief Pain Inventory (BPI) application, which allows assessing pain from a multidimensional perspective (pain intensity and interference with general activities, mood, mobility, work, personal relationships, sleep and enjoyment of life, etc.) (primary outcome), the primary outcome will be the Brief Pain Inventory (BPI) score, which assesses pain levels, sleep quality, mood, fatigue, disability, use of analgesics, etc. Secondary outcomes are the impact of pain on quality of life, depressive symptoms. Predictors of the placebo effect will also be evaluated, through the Verbal Numerical Pain Scale (NPS, 0-10) scores in the last week and through the BPI scores, using a multiple hierarchical model. Among potential predictors, there is disability due to pain, psychological profile, drugs in use. In addition to these, the index of inflammatory markers (serum interleukins IL1-, IL-6, IL-10; TNF-alpha and C-reactive protein); serum levels of endorphins, brain-derived neurotrophic factor (BDNF), S-100B protein and the polymorphisms Val66Met of the BDNF gene and Val158Met of the COMT enzyme gene. Will be included 100 women with FM, randomized to receive active (n=50) or sham (n=50) tDCS, aged between 18 and 65 years. Randomization will be stratified according to the placebo effect response potential, determined after a simulated tDCS session. A variation in NPS (0-10) equal to or greater than 30% after a simulated tDCS session will classify them as high responders to the placebo effect. The follow-up time will be four weeks after a single treatment session. In this way, it is intended to produce consistent evidence for the use of this low-cost technique in the treatment of patients of the Unified Health System, which will be directed to patients with chronic pain at the same time, which will provide data to subsidize the feasibility of studying the effect of this complementary therapy in other conditions, such as refractory depression and neurorehabilitation. In addition, to provide data to better understand tDCS response predictors in outcomes that are related to the impact of pain on the quality of life of conditions that generate a lot of suffering and high costs to the health system.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 65 years; who can read and write, with a confirmed diagnosis of FM according to the American College of Rheumatology criteria (2010-2016). Pain score equal to or greater than six on the Numerical Pain Scale (NPS 0-10) on most days of the last 3 months.

Exclusion Criteria:

* Residing outside the greater Porto Alegre area and pregnancy. Contraindications to TMS and tDCS: metallic implant in the brain; medical devices implanted in the brain, cardiac pacemakers; cochlear implant; history of alcohol or drug abuse in the last 6 months; neurological pathologies; hx of head trauma or neurosurgery; decompensated systemic diseases and chronic inflammatory diseases (lupus, rheumatoid arthritis, Reiter's syndrome); uncompensated hypothyroidism; personal history of cancer, past or undergoing treatment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in pain level - first phase | Time Frame: 1 month
  Change from before and after the First phase of treatment on Pain scores assessed by a Numerical Pain Scale (NPS 0 to 10) (0 means no pain - 10 means the worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No